CLINICAL TRIAL: NCT04959461
Title: A Pilot Trial to Prevent Intoxicated and Impaired Driving Among Adolescents
Brief Title: Preventing Impaired Driving Among Adolescents
Acronym: webCHAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stanford University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Karen Osilla, Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 61874; R34AA027689 (NIH)
Record Dates: First submitted 2021-06-16; First posted 2021-07-13 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Substance-Related Disorders
Keywords: impaired driving
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Teen participants will be randomized to a single-session, self-guided web-intervention called webCHAT or usual care after completing an online baseline survey. Participants will complete follow-up surveys 3 and 6-months after baseline.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- webCHAT (Experimental): Single session 20-40minute self-guided web program that discusses promotes healthy decision making around driving and discusses the risks of alcohol and cannabis-influenced driving.
  Interventions: Behavioral: webCHAT
- Usual Care (Active Comparator): Existing driving school education
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: webCHAT — A self-guided, single session web intervention that utilizes a motivational interviewing style to prevent impaired driving
  Arms: webCHAT
Behavioral: Usual Care — 6 hours of driver education
  Arms: Usual Care

SUMMARY:
The primary goal of this project is to evaluate the efficacy of webCHAT, a single-session web-intervention, on reducing impaired driving among adolescents receiving behind-the-wheel training at driver education programs.

DETAILED DESCRIPTION:
Alcohol and marijuana (AM) are the most commonly used substances among adolescents in the U.S. The consequences of AM use are significantly higher relative to use of either substance alone. This study builds on effective interventions that have demonstrated reductions in alcohol and/or marijuana use and reduced consequences one year later, and proposes to adapt one of those interventions, CHAT, to the web (web-CHAT). The investigators will evaluate the efficacy of web-CHAT among 15.5-17-year-old adolescents (n=150) recruited when teen participants are attending behind-the-wheel training. The study has the potential to promote public welfare by improving adolescent health outcomes and reducing risky driving behaviors that can have substantial monetary and social costs, as well as by providing unique insight into what mediates reduced risky driving attitudes behaviors among those in the intervention. The study is innovative because it is for both youth who are at risk for substance use as well as those who are not, and it is delivered during a teachable moment when adolescents receive driver's education. Finally, this study can provide unique insights about the efficacy of web-CHAT to reduce marijuana initiation, use, and risky driving attitudes in the context of a changing marijuana policy climate. A 3-year study is proposed to test the feasibility of research procedures in a driver education setting and pilot the efficacy of web-CHAT. The investigators will test whether web-CHAT reduces alcohol and/or marijuana initiation or use compared to teens in UC, at three and six-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 15.5-17 year olds enrolled in driver education school
* Access to a computer or smartphone
* Within one month of taking their driver's licensing exam

Exclusion Criteria:

* Under 15.5 or over 17 years old
* Not enrolled in one of the participating schools
* Non-English speaking

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Alcohol and/or Cannabis use (scale from Monitoring the Future survey) | Baseline through month 6
  Number of days of alcohol, marijuana, and/or co-use (concurrent and simultaneous) in the past 30 days

SECONDARY OUTCOMES:
Driving under the influence behaviors (scale from Monitoring the Future survey) | Baseline through month 6
  Number of times they drove a car, motorcycle or other vehicle after using marijuana, alcohol, and/or both in the past 30 days
Passenger driving behavior behaviors (scale from Monitoring the Future survey) | Baseline through month 6
  Number of times they were a passenger in a car or other vehicle with a driver who had beenin the past 30 days drinking alcohol and/or using marijuana

CONTACTS AND LOCATIONS:
Overall Officials: Karen Osilla, PhD, Principal Investigator — Professor
Locations (2):
- United States (2):
  - DriveSafe Driving School, Denver, Colorado
  - DriveSafe Driving School, Dearborn, Michigan

IPD SHARING:
Plan to Share IPD: Yes
Following the NIH Data Sharing Policy and Implementation Guidelines, we plan to make the dataset available for sharing at the time that the main project findings are accepted for publication. That is, the raw data file and codebook, which will initially be used for internal study team purposes, will be available for public use after our main intervention effects paper is published; within one year of the final year of funding.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After our main intervention effects paper is published; within one year of the final year of funding.

REFERENCES:
- [Derived] Osilla KC, D'Amico EJ, Smart R, Rodriguez A, Nameth K, Hummer J. Study design to evaluate a web-intervention to prevent alcohol and cannabis-impaired driving and use among adolescents in driver education. Addict Sci Clin Pract. 2023 Mar 24;18(1):17. doi: 10.1186/s13722-023-00373-2. PMID 36964608